CLINICAL TRIAL: NCT07044466
Title: Real-world Assessment of Social Functioning During OUD Treatment: Integrating Reports From Patients and Their Concerned Significant Others
Brief Title: Social Functioning in Opioid Use Disorder
Acronym: OUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Amber Jarnecke, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00144221
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT4CBT-Buprenorphine (Experimental): CBT4CBT-Buprenorphine
  Interventions: Behavioral: CBT4CBT-Buprenorphine

INTERVENTIONS:
Behavioral: CBT4CBT-Buprenorphine — CBT4CBT-Buprenorphine is an evidence-based, Internet-delivered cognitive behavioral therapy program for individuals prescribed buprenorphine by a medical provider. It includes eight 30-minute modules.

SUMMARY:
Problems with social functioning are core to opioid use disorder (OUD), though specific, modifiable social functioning targets and how they relate to OUD treatment outcomes are poorly understood. This study will utilize both data from both patients with OUD and their concerned significant other (CSO) to examine associations between specific social functioning metrics and OUD treatment outcomes. Findings from this study will inform future precision-medicine approaches for people with OUD, a population in significant need of enhanced treatment approaches to combat opioid morbidity and mortality.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) continues to be associated with high rates of morbidity and mortality and has a significant impact on affected individuals, their families, and their communities. Problems related to social functioning are part of OUD criteria and a wealth of research suggests that individuals with OUD may be prone to experiencing isolation, loneliness, lack of social support, and poor conflict resolution and problem-solving skills in interpersonal contexts. Emerging evidence suggests that OUD treatment, particularly behavioral treatments adjunctive to medications for OUD (MOUD), may improve social functioning and that gains in social functioning may have beneficial impacts on OUD recovery; however, the specific social functioning metrics that are associated with positive OUD treatment trajectories are understudied. Further, much of the extant literature has only examined social functioning from the lens of the patient with OUD, even though reports from concerned significant others (CSOs) may have valuable predictive utility. The proposed study seeks to address gaps in the field by examining how affiliative social engagement behaviors, social reward, and social connection change and are associated with positive OUD treatment outcomes among a sample of 100 patient-CSO dyads. The study will combine established ecological momentary assessment (EMA) methods with the use of an innovative smartwatch-based application (i.e., SocialBit) in a single-armed trial to assess both subjective self-reports and objective measurements of social functioning from patients with OUD and a non-substance using CSO. Aim 1 will determine how patient-reported and CSO-reported social behaviors, social reward, and social connection change during OUD treatment; Aim 2 will identify if patient-reported and CSO-reported social behaviors, social reward, and social connection predict MOUD adherence and opioid craving; Exploratory Aim 3 will validate the use of SocialBit for assessing social connection in an OUD treatment sample. There is an urgent need to address how social functioning contributes to OUD and opioid overdose, and to take a "whole person" approach to treatment. Findings have strong potential to inform future precision-medicine approaches focused on the dual targets of OUD and social functioning.

ELIGIBILITY:
Inclusion Criteria:

* Any sex or gender; any race or ethnicity; aged 18 years or older
* Patient participants must meet DSM-5 diagnostic criteria for current (i.e., past 12 months) OUD (assessed via the Quick Structured Clinical Interview for DSM-5; Quick SCID)
* Patient participants must be on buprenorphine, as prescribed by their provider, for no more than 4 weeks prior to study initiation
* Concurrent substance use disorders (e.g., alcohol, cannabis) for the patient participant are acceptable, provided opioids are the patient participant's primary substance of choice
* Patient participants must identify a CSO participant who consents to participation in the study as well

Exclusion Criteria:

* Moderate-to-severe opioid withdrawal as defined by a score of ≥21 on the Subjective Opioid Withdrawal Scale
* Meeting DSM-5 criteria for a history of or current psychotic or bipolar disorders
* Current suicidal or homicidal ideation and intent; participants who present a serious suicide risk are likely to require hospitalization during the study and they will be referred clinically
* CSO participants meeting DSM-5 criteria for opioid use disorder or any other substance use disorder, excepting tobacco use disorder
* Severe interpersonal violence in the past six months between the patient and the CSO, as defined by an adapted version of the Conflict Tactics Scaled Revised (CTS-2)
* Pregnancy for patient participants
* Prisoners, institutional individuals, and children will not be recruited for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Affiliative social behaviors | Week 1 to Week 14
  Checklist of 12 items assessing social interaction behaviors (adapted from the Social Behavior Inventory; Moskowitz, 1994), summed, averaged, and ipsatized to assess dominant behavior, submissive behavior, agreeable behavior, and quarrelsome behavior. Higher scores reflect greater frequency of the type of behavior.
Social reward | Week 1 to week 14
  1 item assessing how much an individual liked their social interactions (adapted from Geyer, et al., 2018). Higher scores reflect more enjoyment from social interactions.
Social connection | Week 1 to week 14
  1 item assessing how close an individual felt with others (adapted from Flores et al., 2015). Higher scores reflect greater feelings of closeness.
Medication for opioid use disorder adherence | Week 1 to week 14
  2 items assessing daily adherence to taking medication for opioid use disorder (response options: yes; no, I took it, but not as prescribed; no, I did not take buprenorphine) and at what dose (in mgs).
Craving | Week 1 to week 14
  1 item assessing craving for opioids (adapted from Mun et al., 2021; Ellis et al., 2022). Higher scores reflect greater craving.

CONTACTS AND LOCATIONS:
Overall Officials: Amber M Jarnecke, PhD, Principal Investigator — Medical University of South Carolina; Rachel Tomko, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Documentation to be made available will include a study protocol, reference to study publication of primary outcomes, data sets, case report forms, a data dictionary, and study-specific notes. Variables in the NIMH Data Archive (NDA) data dictionary will include a description, variable name, variable label, and standard codes for missing values. Coded interview data, scale composites, recodes will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: A NDA Data Submission Agreement will be signed and a NDA Data Expected section will be completed within six months of receipt of the award. Data will be deposited to NDA every six months, according to the NDA submission deadlines. The research community will have access to the full data set approximately 18 months following the end of the study or after the primary paper has been accepted for publication, whichever happens first. Study data deposited will be available to the research community indefinitely.
Access Criteria: Data will be findable for the research community through NDA.